CLINICAL TRIAL: NCT01706029
Title: Multidimensional Evaluation of Pain in Rheumatoid Arthritis (Douleur PR)
Brief Title: Pain Evaluation in Rheumatoid Arthritis
Acronym: Douleur-PR
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I11013/
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sampling of blood for dosage of IL-6, IL-17 and IL-33 serum level
Oversight: Data Monitoring Committee: No

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory chronic rheumatism where the pain remains the priority domain of improvement for the patients instead a good control of the inflammatory disease by treatments, even biotherapeutics .

Some studies show that less than 50 % of the patients is satisfied by the care of the pain, whereas the criteria of evaluation of the RA improve under treatment. The chronic pain, is a complex and multifactorial subjective phenomenon requiring a multidimensional evaluation, while the current criteria of follow-up of the RA (DAS28, ACR criteria) investigate the pain in a single dimension that is the pain intensity.

So, the investigators do not arrange explanation for this observed dichotomy between the improvement of the clinical and biological inflammatory criteria of the RA and on the other hand the persistence of pain.

On the other hand, the interleukin (IL)-6, IL-17 and IL-33 are cytokines occurring in the physiopathology of RA and probably in the pain processing according to recent data of the literature.

The aim of this study is:

* to assess the multidimensional origin of the pain in RA patients by means of questionnaires
* to look for a possible correlation between the serum level of cytokines and pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults with RA treated with DMARDs and/or biotherapy,
* Capable of providing written consent

Exclusion Criteria:

* Patients affected by a painful disease other one than RA,
* Fibromyalgia,
* A malignancy disease,
* An hemopathy,
* Psychiatric disorders or dementia and
* Acute infectious diseases and
* Receive or had received anti-IL6 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected from those coming to the Department of Rheumatology of each partcipating center.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pain | At day 1
  Multidimensional evaluation of the pain using standard questionnaires: HAS, Beck and Speilberger , Erosion Narrow Score and Fibromyalgia diagnostic criteria

SECONDARY OUTCOMES:
Patients pain care | At day 1
  Estimate the satisfaction of the patients towards the coverage (care) of their pain by means of VAS and verbal scale of satisfaction
Correlation | At day 1
  Estimate the correlation between the activity of the RA and the multidimensional evaluation of pain using DAS28 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Vergne-Salle, MD, Principal Investigator — CHU Limoges
Locations (7):
- France (7):
  - CHU Bordeaux- Pellegrin, Bordeaux
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Hôpital R. Salengro, Lille
  - Service de Rhumatologie, Limoges
  - CHU Hôtel-Dieu, Paris
  - CHU Bois-Guillaume, Rouen
  - CHU Hautepierre, Strasbourg